CLINICAL TRIAL: NCT04491539
Title: Adapting the Finding Respect and Ending Stigma Around HIV (FRESH) Intervention for the Dominican Republic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Henna Budhwani, Professor, Florida State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 526497; 5R21TW011761-02 (NIH)
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Hiv
Keywords: Stigma; Intervention; HIV; Dominican Republic; Spanish
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Intervention Model Description: Pre- and post- intervention participation assessment; arms represent participant types, either healthcare worker or person with HIV (PWH) client.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare Workers or Providers (Experimental): Healthcare Workers or Providers receiving the FRESH intervention. Arm to test the intervention's effect on this specific population.
  Interventions: Behavioral: Finding Respect and Ending Stigma around HIV (FRESH)
- Clients (Experimental): People with HIV Clients receiving the FRESH intervention. Arm to test the intervention's effect on this specific population.
  Interventions: Behavioral: Finding Respect and Ending Stigma around HIV (FRESH)

INTERVENTIONS:
Behavioral: Finding Respect and Ending Stigma around HIV (FRESH) — The Finding Respect and Ending Stigma around HIV (FRESH) intervention is theoretically informed by Social Cognitive Theory (SCT) and Interpersonal Contact theory (ICT) and was specifically designed for delivery in high-stigma settings, such as Dominican Republic. FRESH was originally developed in Africa to address HIV-related stigma, and later was adapted to address intersectional stigmas experienced by sexual and gender minorities (SGM) living with HIV in the United States Deep South. To our knowledge, FRESH will be the first intervention to address intersectional stigmas experienced by men who have sex with men, transgender women, and people living with HIV in clinical settings in the Spanish-speaking Caribbean.

SUMMARY:
This research has the potential to make important contributions toward HIV and intersectional stigma reduction across the Spanish-speaking Caribbean. It will do so by adapting and testing a patient-provider, clinic-based intersectional stigma-reduction intervention -- Finding Respect and Ending Stigma around HIV (FRESH) -- for the Dominican Republic. Preliminary results from this R21 study (e.g. workshop satisfaction, stigma outcomes, HIV continuum of care outcomes, etc.) will inform the development of an investigator-initiated R01 proposal to conduct a full scale randomized controlled trial of the adapted FRESH intervention.

DETAILED DESCRIPTION:
The proposed study addresses the high level of stigma against people living with HIV (PLWH), particularly gender and sexual minorities, that is embedded in the Dominican Republic's HIV treatment system through the adaptation and testing of a patient-provider intervention -- Finding Respect and Ending Stigma around HIV (FRESH). The Dominican Republic is a high priority setting with an increasing need for HIV stigma reduction studies. The Caribbean holds the second highest regional burden of HIV in the world, yet receives insufficient HIV-related stigma research funding. The Dominican Republic is 1 of 5 countries that accounts for over 95% of all Caribbean HIV infections; it also has a significant concentrated HIV epidemic, a deeply conservative society in which PLWH are stigmatized, and an exceptionally low national viral load suppression rate. To accomplish this pilot study, three Specific Aims are proposed. Aim 1 is to explore sources, characteristics, and consequences of HIV-related and intersectional stigmas experienced in healthcare settings to inform the adaptation of FRESH. To accomplish Aim 1, we will conduct qualitative in-depth interviews with healthcare workers who provide HIV care, focus groups with MSM, and in-depth interviews with trans- women. Aim 2 is to adapt FRESH to address stigmas experienced these individuals in the Dominican Republic. We will apply the Aim 1 findings using the ADAPT-ITT framework to systematically adapt FRESH, an intervention that has been employed to reduce stigma in healthcare settings in Africa and the United States. Through an iterative process, each revision of FRESH will be shared with both PLWH and healthcare workers to solicit and incorporate their feedback about each version of the adapted intervention. Aim 3 will pilot-test the adapted intervention to obtain estimates of its ability to reduce stigmatizing attitudes and behaviors from HWs and experiences of stigma reported by sexual and gender minorities (SGM) and non-SGM clients living with HIV (primary); while exploring if FRESH has the potential to influence clinic-level outcomes. By adapting and testing the FRESH intervention for the Spanish-speaking Caribbean, FRESH could become a validated, multi-region HIV and intersectional stigma reduction intervention designed specifically for healthcare settings in high-stigma, culturally conservative, resource-constrained communities; such a scientific development would be a significant contribution to HIV stigma reduction efforts in the Caribbean and globally.

ELIGIBILITY:
Inclusion Criteria for health worker participants:

* Minimally 18 years and 0 months of age
* Works at one of the three study sites
* Interacts with people living with HIV
* Spanish speaking
* Can read Spanish text
* Able and willing to provide informed consent

Inclusion Criteria for people living with HIV participants:

* Minimally 16 years and 0 months of age
* Is HIV-positive
* Spanish speaking
* Receives treatment at one of the three study sites
* Identifies as an SGM
* Able and willing to provide informed consent

Exclusion Criteria:

• Does not meet inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All data gathered during the proposed study will be available to all participating investigators and institutions. This includes the University of Alabama at Birmingham (UAB), Universidad Iberoamericana (UNIBE), and the Caribbean Vulnerable Communities Coalition (CVC).

REFERENCES:
- [Derived] Budhwani H, Yigit I, Paulino-Ramirez R, Waters J, Bond CL, Varas-Diaz N, Naar S, Nyblade L, Turan JM. Finding Respect and Ending Stigma around HIV (FRESH) intervention in the Dominican Republic: results from a pilot study. BMC Glob Public Health. 2025 Nov 7;3(1):99. doi: 10.1186/s44263-025-00219-w. PMID 41199402
- [Derived] Yigit I, Paulino-Ramirez R, Waters J, Turan JM, Budhwani H. Disclosure concerns moderate the association between internalized stigma and antiretroviral medication adherence among people with HIV in the Dominican Republic. AIDS Care. 2025 Nov;37(11):1950-1958. doi: 10.1080/09540121.2025.2562253. Epub 2025 Sep 24. PMID 40988523

RESULTS

PARTICIPANT FLOW:
Groups:
- Providers or Healthcare Workers: Half the providers received the Finding Respect and Ending Stigma around HIV (FRESH) intervention first, and then 6-months later, the other half of providers received the intervention. The goal of this pilot study was not to compare outcomes by site or intervention receipt order, rather it was to assess the impact of the intervention on each group, in the case providers; thus, we conducted pre- and post-intervention evaluations by participant type.
- People With HIV (PWH) Clients: Half the PWH clients received the Finding Respect and Ending Stigma around HIV (FRESH) intervention first, and then 6-months later, the other half of PWH clients received the intervention. The goal of this pilot study was not to compare outcomes by site or intervention receipt order, rather it was to assess the impact of the intervention on each group, in the case PWH clients; thus, we conducted pre- and post-intervention evaluations by participant type.
Period: Overall Study
Arm/Group | Providers or Healthcare Workers | People With HIV (PWH) Clients
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Providers: Healthcare providers from both clinics that received the FRESH intervention.
- Clients: People with HIV clients from both clinics that received the FRESH intervention.
- Total: Total of all reporting groups
Arm/Group | Providers | Clients | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Customized [Mean (Standard Deviation); unit: years] | 40.40 (10.33) | 32.47 (6.78) | 36.88 (5.61)
Sex/Gender, Customized [Number; unit: participants]
  Male | 4 | 13 | 17
  Female | 16 | 0 | 16
  Not Reported or Other | 0 | 3 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 4 | 6 | 10
  White | 2 | 0 | 2
  Multiracial | 14 | 8 | 22
  Other or Not Reported | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: HIV-related Stigma
Description: For providers, the results are reported for the Opinions about People with HIV sub-scale from the HIV-related stigma among health facility staff scale, 6 questions. Response options are Strongly Agree, Agree, Disagree, and Strongly Disagree. This scale does not include reverse coding. Higher scores indicate higher levels of stigma. The score can range from 5 (min) to 20 (max). For clients, the results are reported for the Experiencing HIV-related Stigma in Healthcare Settings scale, 5 questions. Response options are Never, Rarely, Sometimes, Usually, and Always. This scale does not include reverse coding. Higher scores indicate higher levels of stigma. The score can range from 0 (min) to 20 (max).
Time Frame: Year 2
Population: Pre -and post- survey measures were then compared to assess the change after the FRESH workshop intervention using paired t-tests if the normality was confirmed. The significance level was identified as p<0.05. All analyses were performed with SAS (Version 9.4, Cray, North Carolina, USA).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Providers: Change in scores among providers pre- and post- attending the intervention, regardless of if they received the intervention in the first or second cycle of delivery.
- Clients: Change in scores among people with HIV (PWH) clients pre- and post- attending the intervention, regardless of if they received the intervention in the first or second cycle of delivery.
Arm/Group | Providers | Clients
Number analyzed (Participants) | 20 | 16
units on a scale
  Pre-Intervention | 8.74 (3.12) | 10.25 (3.91)
  Post-Intervention | 7.16 (2.40) | 8.42 (4.03)

2. Primary Outcome: HIV Knowledge Index
Description: Results are reported for the HIV Knowledge Index from providers only. This is not a validated scale but was being tested in the context of this study. It included 13 homegrown questions. Range was 0 (min) to 13 (max), with higher scores indicating greater knowledge.
Time Frame: Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Providers or Healthcare Workers: Change in scores among providers pre- and post- attending the intervention, regardless of if they received the intervention in the first or second cycle of delivery.
- People With HIV (PWH) Clients: Change in scores among clients pre- and post- attending the intervention, regardless of if they received the intervention in the first or second cycle of delivery.
Arm/Group | Providers or Healthcare Workers | People With HIV (PWH) Clients
Number analyzed (Participants) | 20 | 0
units on a scale
  Pre-Intervention | 7.00 (0.58) |
  Post-Intervention | 6.63 (0.76) |

3. Primary Outcome: Empathy and Avoidance in Treating Patients Living With HIV/AIDS
Description: For providers, the results are reported for empathy and avoidance in treating patients living with HIV/AIDS, 11 questions. Response options are Strongly Agree, Agree, Neutral, Disagree, and Strongly Disagree. This scale includes reverse coding. Higher scores indicate higher levels of stigma. The score can range from 11 (min) to 55 (max).
Time Frame: Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Providers or Healthcare Workers | People With HIV (PWH) Clients
Number analyzed (Participants) | 20 | 0
units on a scale
  Pre-Intervention | 37.10 (4.64) |
  Post-Intervention | 38.00 (5.70) |

4. Secondary Outcome: Multiple Discrimination Scale - Orientation
Description: For clients, the results are reported for experiences of discrimination related to sexual orientation, 10 questions. Response options are Yes and No. Higher scores indicate higher levels of stigma. The score can range from 0 (min) to 10 (max).
Time Frame: Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Providers or Healthcare Workers | People With HIV (PWH) Clients
Number analyzed (Participants) | 0 | 16
units on a scale
  Pre-Intervention |  | 0.83 (2.29)
  Post-Intervention |  | 1.45 (2.42)

ADVERSE EVENTS:
Time Frame: Participants were actively monitored over the duration of the 2.5 day intervention but could report adverse events up to 6 months after receipt of the intervention.
Description: No deviation from the clinicaltrials.gov definition.
Groups:
- Providers or Healthcare Workers: Providers received the adapted Finding Respect and Ending Stigma around HIV (FRESH) intervention.
- People With HIV (PWH) Clients: Clients received the adapted Finding Respect and Ending Stigma around HIV (FRESH) intervention.
Arm/Group | Providers or Healthcare Workers | People With HIV (PWH) Clients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16

LIMITATIONS AND CAVEATS:
Data was collected from two clinics and the sample size was small. A selection bias could have affected results wherein providers who were amenable to change may have been more likely to participate and clients with higher levels of self-efficacy may have been more likely to attend the workshop.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04491539/Prot_SAP_000.pdf